CLINICAL TRIAL: NCT03148938
Title: " Digitalization of Neurofunctional Tests Via a Mobile Application, Digital Assessment Multiple Sclerosis (DAMS), for Multiple Sclerosis Patients"
Brief Title: Digitalization of Neurofunctional Tests Via a Mobile Application DAMS for Multiple Sclerosis Patients
Acronym: MSCopilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: P005
Record Dates: First submitted 2017-05-05; First posted 2017-05-11 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-07

CONDITIONS: Multiple Sclerosis
Keywords: DAM; multiple sclerosis; MSFC; application; mobile
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Patients will perform one or two visits at 15 days interval. Healthy volunteers will only perform one visit. Patients and healthy volunteers will be randomly assigned to either traditional/digital group (Group A) or digital/traditional group (Group B), followed by a crossover to the other group at day 15 for patients who will do two visits.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Multiple Sclerosis (Experimental): Patients will perform one or two visits at 15 days interval. Patients will be randomly assigned to either traditional/digital group (Group A) or digital/traditional group (Group B), followed by a crossover to the other group at day 15 for patients who will do two visits.
  Interventions: Other: Digital Assessment on mobile
- Healthy volunteer (Active Comparator): Healthy volunteers will only perform one visit. Healthy volunteers will be randomly assigned to either traditional/digital group (Group A) or digital/traditional group (Group B).
  Interventions: Other: Digital Assessment on mobile

INTERVENTIONS:
Other: Digital Assessment on mobile — The digital assessment is composed on 4 tests:
  * walking test
  * coordination test
  * attention test
  * vision test

SUMMARY:
Multiple Sclerosis (MS) is a chronic immune-mediated inflammatory disease with a broad diversity of symptoms and fluctuating progression patterns. Clinical assessments are challenging and are continually reviewed and enhanced. Optimal multiple sclerosis care depends on early detection of disease progression. The Digital self-Assessment for Multiple sclerosis (DAM) mobile program was developed by Ad Scientiam in order to create a robust and clinically validated remote monitoring platform for MS patients and clinicians. The correlation between DAM version 0 (the first iteration of DAMS) and Multiple Sclerosis Functional Composite (MSFC) has been clinically evaluated in a preliminary study in 30 subjects. DAM version 0 and MFSC global scores were correlated. However, the cognition test had a poor reproducibility and clinicians expressed the wish to measure a walking range rather than a walking speed. Even though vision is the main sense impacting all other tests, particularly when interacting with a mobile, visual tests are rarely performed in real life. A new version of DAM version 0, DAMS, was therefore developed with the addition of the Sloan Low Contrast Letter Acuity Test (SLCLAT), the replacement of the walking speed test with a walking distance test and the Paced Auditory Serial Addition Test (PASAT) by a new version of the cognitive test which resembles the Symbol Digit Modalities Test (SDMT).

The hypothesis is that systematic and prospective multi-dimensional data collection of MS disabilities through the DAMS mobile application will refine the quality and accuracy of both clinicians and patients' knowledge of the disease progression and will ultimately improve the current care of patients.

To test this assumption, the statistician will analyze:

1. The global diagnostic performance of DAMS with (DAMS 4 tests) and without (DAMS 3 tests) the low contrast vision test versus standard MS scales
2. The test-retest reliability of DAMS' scores at a 15 day interval

ELIGIBILITY:
Inclusion Criteria:

MS patients:

* subjects: 18 Years to 60 Years
* with a confirmed and documented MS diagnosis, per the 2010 Revised McDonald criteria
* with or without MS maintenance and/or symptomatic treatment, if MS maintenance and/or symptomatic treatment: stable for the past 6 months before enrolment (Centrally acting antalgics, antidepressant or neuroleptic treatment are authorized but shall not be modified in the past 2 months before enrolment)
* with an EDSS [0;7] in the past 6 months before enrolment
* with an EDSS [0;7] in the past 6 months before enrolment
* with no evidence of EDSS score change since the last measure available
* with no evidence of relapse in the past 6 months before enrolment
* enrolled in or benefiting of a Social Security program
* who have read the information sheet and signed the informed consent form

Healthy volunteers:

* subjects: 18 Years to 60 Years
* with no evidence of walk limitation (as per clinician's judgment) nor walking aid
* no personal and familial history of inflammatory disease (e.g. rheumatoid arthritis) or multiple sclerosis
* matched to the sociodemographic characteristics of MS patients sample (age, sex, height, weight, education)
* enrolled in or benefiting of a Social Security program
* who have read the information sheet and signed the informed consent form

Non-Inclusion Criteria:

MS patients and Healthy volunteers:

* Participants wearing pacemakers, implantable defibrillators, or hearing aids
* Inability to use their right hand for the Coordination test (MCT)
* Evidence of neurologic or psychiatric disorder other than MS, including but not limited to major head trauma, seizures or systemic medical diseases that are likely to affect cognitive functioning
* Evolutive rheumatology disease
* Any vision (ex. short-sightedness (-6; +6); congenital dyschromatopsia and glaucoma) or hearing conditions that could influence the performing of the tests
* Omission of the usual visual and/or walking aids if it's usually needed
* Acute asthenia (score>7 on a visual analogic scale)
* Systemic corticosteroid treatment in the past 30 days before enrolment
* Intramuscular botulinic toxin injection in the past 4 months before enrolment
* Change in centrally acting antalgic, antidepressant or neuroleptic treatment in the past 2 months before enrolment
* Rehabilitation in the past 6 months before enrolment
* Pregnant and nursing women - Person under guardianship or curatorship
* Bedridden patients or patients with a daily activity of less than 2 hours per day
* Inability to use a mobile application
* Current drugs or/and alcohol abuse that could influence performance on the tests (clinician's judgment)
* Participation to another study Healthy volunteers who will not match the sociodemographic characteristics of MS patients will not be included in the study.

Exclusion Criteria:

* Patient experiencing a relapse once enrolled in the study
* Patient with a maintenance and symptomatic MS treatment modification
* Use of centrally acting antalgics, antidepressant or neuroleptic once enrolled in the study
* Substance or/and alcohol abuse that could influence performance on the tests between inclusion and follow-up visits (clinician's judgement)
* Omission or change in the usual visual and/or walking aids
* Acute asthenia (score>7 on a visual analogic scale) at the follow-up visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of DAMS 3 test measured with digital assessment versus MSFC measured with traditional tests. | Day 0
  Determine the diagnostic performance of DAMS 3 tests (not included the vision test results) for the detection of MS patients in a population of healthy volunteers and MS patients (with Expanded Disability Status Scale (EDDSS) score [0;7]) compared to the traditional tests (MSFC)

SECONDARY OUTCOMES:
Diagnostic performance of DAMS 4 tests measured with digital assessment versus MSFC (with vision test) measured with traditional tests | Day 0
  Determine the diagnostic performance of DAMS 4 tests (included the vision test results) for the detection of MS patients in a population of healthy volunteers and MS patients (with Expanded Disability Status Scale (EDSS) score [0;7]) compared to the conventional MSFC + Sloan low contrast letter acuity test
Diagnostic performance of DAMS 3 tests measured with digital assessment versus MSFC revised measured with traditional tests | Day 0
  Determine the diagnostic performance of DAMS 3 tests for the detection of MS patients in a population of healthy volunteers and MS patients (with EDSS score [0;7]) compared to a revised form of MSFC in which PASAT has been replaced by SDMT
Diagnostic performance of DAMS 4 test measured with digital assessment versus MSFC revised with vision test measured with traditional tests | Day 0
  Determine the diagnostic performance of DAMS 4 tests for the detection of MS patients in a population of healthy volunteers and MS patients (with EDSS score [0;7]) compared to a revised form of MSFC in which PASAT has been replaced by SDMT and SLCLAT added.
Correlation between DAMS 3 tests measured with digital assessment and MSFC measured with traditional tests | Day 0
  To assess correlation between DAMS 3 tests and MSFC in MS patients and healthy volunteers
Correlation between DAMS 3 tests measured with digital assessment and MSFC revised measured with traditional tests | Day 0
  To assess correlation between DAMS 3 tests and MSFC in which PASAT has been replaced by SDMT in MS patients and healthy volunteers
Correlation between DAMS 4 tests measured with digital assessment and MSFC with vision test measured with traditional tests | Day 0
  To assess correlation between DAMS 4 tests and MSFC with vision test result in MS patients and healthy volunteers
Correlation between DAMS 3 tests measured with digital assessment and MSFC revised with vision test measured with traditional tests | Day 0
  o assess correlation between DAMS 3 tests and MSFC in which PASAT has been replaced by SDMT with vision test result in MS patients and healthy volunteers
Compare scores of digital assessment versus scores of traditional tests | Day 0
  To compare the scores obtained with each DAMS' evaluation test [mobile walking test, coordination test, attention test, vision test ] to those obtained with traditional tests (T25FW, 9-HPT, PASAT, SDMT, SLCLAT) in MS patients and healthy volunteers
Compare scores of digital assessment at day 0 versus 15 days later | Day 15
  To assess the test-retest reliability of DAMS 3 and 4 tests during the study in MS patients with EDSS score [0;7]
Safety of Mobile assessment with the collect of all the adverse events | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth MAILLART, MD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (10):
- France (10):
  - Hôpital le Bocage, Dijon
  - Hôpital Saint-Phllibert, Lille
  - Hôpital La Timone Adulte, Marseille
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Pasteur, Nice
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Maison Blanche, Reims
  - Hôpital Saint Hélier, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Hautepierre, Strasbourg